CLINICAL TRIAL: NCT00129272
Title: Stress Response and Smoking Cessation in Depressed Youth
Brief Title: Effectiveness of Bupropion for Treating Nicotine Dependence in Young People
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Uma Rao, Professor of Psychiatry, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-15131-1
Record Dates: First submitted 2005-08-04; First posted 2005-08-11 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Tobacco Use Cessation; Tobacco Use Disorder
Keywords: adolescents, cigarettes, smoking, tobacco
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use Disorder; Smoking | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupropion (Wellbutrin-SR) (Active Comparator): Using a double-blind, randomized, placebo-controlled design, smokers received active treatment with Bupropion-SR (150 mg. twice daily) in conjunction with cognitive-behavior therapy (weekly sessions) for smoking cessation over a 9-week period.
  Interventions: Drug: Bupropion-SR
- Matching Placebo (Placebo Comparator): Using a double-blind, randomized, placebo-controlled design, smokers received treatment with a matching placebo (to Bupropion-SR 150 mg) twice daily in conjunction with cognitive-behavior therapy (weekly sessions) for smoking cessation over a 9-week period.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bupropion-SR — 150mg tablets taken orally twice daily for 9 weeks.
  Other Names: Wellbutrin-SR
  Arms: Bupropion (Wellbutrin-SR)
Other: Placebo — Matching placebo (to Buproion-SR) twice daily for 9 weeks.
  Other Names: Placebo match for Bupropion (Wellbutrin) SR
  Arms: Matching Placebo

SUMMARY:
Little is known about the best ways to help young people stop smoking. Bupropion (a medication marketed as Wellbutrin or Zyban) has proved helpful in treating adult smokers. The purpose of this study is to determine if bupropion is also effective in treating smokers between the ages of 12 and 25 years old. This study also compares the effectiveness of bupropion used as a supplement to behavioral treatment versus behavioral treatment used alone. In addition, the study evaluates whether hormonal response to stress measured prior to the start of treatment predicts whether individuals respond well to treatment with medication.

DETAILED DESCRIPTION:
Cigarette smoking and other forms of tobacco exposure are one of the leading preventable causes of morbidity and mortality in the United States. Most smokers begin smoking during adolescence, and though they seem motivated to quit smoking, they frequently fail. Although behavioral treatments are available, they have not been very successful in past studies.

Depressed adults may have more difficulty quitting smoking than non depressed adults; this finding may also apply to depressed youth. The purpose of this study is to determine the effectiveness of bupropion in combination with standard behavioral treatment in helping young smokers quit, as compared to behavioral treatment alone. Finally, the study examines whether hormonal response to stress measured prior to treatment initiation predicts whether individuals respond well to treatment with bupropion.

Participants in this double-blind study will be randomly assigned to receive either bupropion or placebo. Both groups will receive behavioral treatment. The trial will last for 9 weeks, with weekly study visits. Study visits will last 30 minutes to 1 hour and will include medication monitoring, self-reported and biological measures of smoking, and behavioral treatment. Participants will have follow-up visits six months after completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has smoked at least 10 cigarettes each day for 3 or more months
* Weighs at least 90 lbs
* Motivated to quit smoking and has had at least one previous failed attempt
* Speaks, reads, and writes English
* Either diagnosed as depressed OR no history of a psychiatric disorder

Exclusion Criteria:

* History of bipolar disorder, eating disorder, schizophrenia, schizoaffective disorder, autism, or non-nicotine substance use disorder in the 6 months prior to study entry
* Currently suicidal or with a history of a suicide attempt in the 6 months prior to study entry
* Psychotic symptoms
* Use of psychotropic medication(s)
* Serious medical condition
* Prior use of bupropion for smoking cessation
* Currently using other smoking cessation treatments

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 172 (Actual)
Dates: Start 2004-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uma Rao, MD, Principal Investigator — University of Texas Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants between ages 12 and 25 years who smoked at least 10 cigarettes per day over a period of 6 months were recruited between 2004 and 2010 through advertisements in local newspapers and flyers in local community agencies and primary care clinics.
Pre-assignment Details: Participants completed an assessment for nicotine dependence and psychiatric disorders, and a laboratory stress study to assess baseline salivary cortisol over 2 hours and cortisol responses to a psychosocial stressor (public speaking and arithmetic tasks). Those who continued to meet study criteria were then randomized to active drug or placebo.
Groups:
- Active Drug (Burpropion-SR): In total 172 participants were recruited, and 144 were randomized.
  Using a double-blind, randomized, placebo-controlled design, participants were randomized to active drug or placebo using the modified Efron's biased coin toss method to ensure that the drug/placebo cells are balanced with respect to severe depression, presence of nicotine dependence symptoms and gender.
  Participants received active treatment with Bupropion-SR (150 mg. twice daily) in conjunction with cognitive-behavior therapy (weekly sessions) for smoking cessation over a 9-week period.
  The participants had weekly visits with the target quitting date set for Day 8. The medication checks lasted about 30-45 minutes. The focus was on elicitation of smoking status, nicotine craving and withdrawal symptoms, depressive symptoms and side effects. Body weight and vital signs were measured as well as expired air for CO and urine cotinine levels. Plasma drug levels were obtained at 5 and 9 weeks of treatment.
- Matching Placebo: This arm included placebo treatment twice daily for 9 weeks. Drug and placebo were compounded to look identical, masking both drug type and dosage.
  All participants (both drug and placebo groups) received a modified version of the brief office intervention program for adolescent smokers, developed by the American Medical Association. Subjects met with a research counselor for 10 consecutive weekly sessions. The initial session (baseline visit) was 60 min. while the remaining sessions were 20-30 min. Each session was individualized to the needs of the adolescent, based on information gathered at the baseline assessment. The brief office intervention materials include checklists and guidelines for each session to assist the counselor in tailoring the session to the needs of the youth. It involved motivational interviewing, incorporating stages of change, peer and parental and other social influences; negative affect and other psychological factors, addiction and self-efficacy.
Period: Overall Study
Arm/Group | Active Drug (Burpropion-SR) | Matching Placebo
Started | 71 | 73
Completed | 54 | 51
Not Completed | 17 | 22
Not completed — Lost to Follow-up | 12 | 11
Not completed — Withdrawal by Subject | 5 | 11

BASELINE CHARACTERISTICS:
Groups:
- Active Drug (Bupropion-SR): Using a double-blind, randomized, placebo-controlled design, smokers received active treatment with Bupropion-Sr (150 mg. twice daily) in conjunction with cognitive-behavior therapy (weekly sessions) for smoking cessation over a 9-week period.
  Bupropion-SR: 150mg tablets taken orally twice daily for 9 weeks.
- Total: Total of all reporting groups
Arm/Group | Active Drug (Bupropion-SR) | Matching Placebo | Total
Number analyzed (Participants) | 71 | 73 | 144
Age, Continuous [Mean (Standard Deviation); unit: Years] — Participants were between 12 and 25 years of age.
  Years | 19.6 (3.2) | 18.3 (3.9) | 19.0 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 77
  Male | 33 | 34 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black : non-Hispanic | 9 | 10 | 19
  Black : Hispanic | 0 | 0 | 0
  White : non-Hispanic | 52 | 51 | 103
  White : Hispanic | 0 | 0 | 0
  More than one race : non-Hispanic | 0 | 0 | 0
  More than one race : Hispanic | 10 | 12 | 22
Region of Enrollment [Number; unit: participants] — The data were collected in Southwestern Region of the United States
  participants
    United States | 71 | 73 | 144
Daily smoking diary [Mean (Standard Deviation); unit: cigarettes/day in previous week] — Number of cigarettes smoked per day
  cigarettes/day in previous week | 17.5 (7.6) | 16.4 (6.8) | 16.9 (7.2)
Withdrawal symptoms [Mean (Standard Deviation); unit: units on a scale;range 0-36;higher worse] — Hughes-Hatsukami Withdrawal Scale
  units on a scale;range 0-36;higher worse | 4.3 (3.3) | 4.1 (3.5) | 4.2 (3.5)
Nicotine dependence [Mean (Standard Deviation); unit: units on a scale;range 0-9;higher worse] — Fagerstrom Tolerance Questionnaire
  units on a scale;range 0-9;higher worse | 5.6 (1.6) | 5.4 (1.3) | 5.5 (1.5)
Expired carbon monoxide [Mean (Standard Deviation); unit: Parts per million; higher worse] | 13.9 (5.3) | 14.0 (8.9) | 13.9 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Smoking Behavior
Description: Number of cigarettes smoked daily in the previous week
Time Frame: Nine weeks
Population: Analyzed all randomized participants with last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: cigarettes/day in the previous week
Arm/Group | Active Drug (Bupropion-SR) | Matching Placebo
Number analyzed (Participants) | 71 | 73
cigarettes/day in the previous week | 6.4 (4.3) | 8.9 (5.4)

2. Secondary Outcome: Withdrawal Symptoms
Description: Hughes-Hatsukami Withdrawal Scale
Time Frame: Nine weeks
Population: Analyzed all participants with last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale;range0-36;higher worse
Arm/Group | Active Drug (Bupropion-SR) | Matching Placebo
Number analyzed (Participants) | 71 | 73
units on a scale;range0-36;higher worse | 2.5 (3.3) | 3.1 (4.3)

ADVERSE EVENTS:
Time Frame: Time frame for adverse events was over 9 weeks of treatment.
Description: Adverse events were recorded based on Hughes-Hatsukami Withdrawal Scale and Side Effects Form.
Arm/Group | Active Drug (Bupropion-SR) | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/73
Other Adverse Events (participants affected / at risk) | 7/71 | 8/73
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Drug (Bupropion-SR) (N=71) | Matching Placebo (N=73)
Nausea (Gastrointestinal disorders) | 7 (23) | 6 (16)
Negative affect (Psychiatric disorders) | 3 (5) | 8 (23) — negative mood/affect reported during the course of treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No